CLINICAL TRIAL: NCT05568394
Title: Effects of Manual Therapy Combined With Therapeutic Exercise on Brain Biomarkers in Patients With Chronic Nonspecific Neck Pain: Study Protocol for a Randomized Controlled Trial.
Brief Title: Effects of Manual Therapy Combined With Therapeutic Exercise on Brain Biomarkers in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Sureeporn Uthaikhup, Principal Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-65 2301484
Record Dates: First submitted 2022-10-04; First posted 2022-10-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Neck Pain
Keywords: Neck pain; Manual therapy; Exercise; Magnetic resonance imaging; Magnetic resonance spectroscopy
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A single-blinded design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Manual therapy and therapeutic exercise
  Interventions: Other: Manual therapy combinded with therapeutic exercise
- Control group (Experimental): Routine physical therapy
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Manual therapy combinded with therapeutic exercise — The treatment includes cervical mobilization and specific therapeutic exercises: craniocervical and cervical flexors and extensors, axioscapular muscles, and postural correction (30-40 minutes).
  The participants will attend 20 individual treatment sessions (2 visits per week for 10 weeks).
  Arms: Intervention group
Other: Routine physical therapy — The treatment includes routine physical therapy (e.g., modalities, range of motion and/or gentle stretching exercise) (30-40 minutes).
  The participants will attend 20 individual treatment sessions (2 visits per week for 10 weeks).
  Arms: Control group

SUMMARY:
Structural brain alterations in pain-related areas have been demonstrated in patients with nonspecific neck pain. While manual therapy combined with therapeutic exercise is an effective management for neck pain, its underlying mechanisms are poorly understood. The primary objective of this trial is to investigate the effects of manual therapy combined with therapeutic exercise on brain imaging biomarkers in patients with chronic nonspecific neck pain. The secondary objectives are to assess neurochemical biomarkers, clinical features of neck pain, cervical range of motion and cervical muscle strength.

DETAILED DESCRIPTION:
This study is a single-blinded, randomized controlled trial. Forty-eight participants with chronic nonspecific neck pain will be recruited into the study. Participants will be randomly allocated to either an intervention or control group (1:1 ratio). Participants in the intervention group will receive manual therapy combined with therapeutic exercise for 10 weeks (2 visits per week). The control group will receive routine physical therapy. Primary outcomes are brain imaging biomarkers (cortical gray matter: volume, thickness and area, and white matter: fractional anisotropy and mean diffusivity) in pain-related areas. Secondary outcomes are neurochemical biomarkers (N-acetylaspartate, NAA; creatine, Cr; glutamic acid/glutamine, Glu/Gln; myoinositol, mI; and choline, cho), clinical features (neck pain intensity, duration, neck disability and psychological symptoms), cervical range of motion and cervical muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* a history of nonspecific neck pain for ≥ 3 months
* an average pain intensity over the past week ≥ 35 mm. on a visual analogue scale (VAS)

Exclusion Criteria:

* a history of head and neck injury or surgery
* known or suspected vestibular pathology or dizziness caused by underlying pathology in the ear, brain and sensory nerve pathways (e.g. benign paroxysmal positional vertigo) and/or vascular disorders
* any neurological or musculoskeletal condition that could affect the outcomes (e.g., scoliosis, torticollis, myofascial pain syndrome, fibromyalgia and rheumatoid arthritis)
* metabolic conditions (e.g., diabetes, obesity (BMI > 30 kg/m2) and hypertension)
* psychological symptoms (e.g., anxiety, depression and schizophrenia)
* contraindications to MRI (e.g., pregnancy/breastfeeding, claustrophobia and ferromagnetic implants)
* receiving physiotherapy treatment for their neck conditions in the past 12 months.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Cortical gray matter: volume and thickness | At baseline and post-intervention
  Cortical gray matter (volume and thickness) will be measured in pain-related areas (thalamus, prefrontal cortex (PFC), primary somatosensory cortex (S1), primary motor cortex (M1), insula, cingulate cortex, precuneus, temporal lobe and periaqueductal gray matter) using a Magnetic resonance imaging (MRI) machine

SECONDARY OUTCOMES:
Neurochemical biomarkers: N-acetylaspartate (NAA), creatine (Cr), glutamic acid/glutamine (Glu/Gln), myoinositol (mI), and choline (cho) | At baseline and post-intervention
  Neurochemistry biomarkers will be measured using single-voxel proton magnetic resonance spectroscopy (1H-MRS) in dorsolateral prefrontal cortex (DLPFC), primary somatosensory cortex (S1), anterior cingulate (ACC), insula and thalamus.
Neck pain intensity | At baseline and post-intervention
  The average intensity of neck pain will be assessed by using a 0-10 cm visual analogue scale (VAS), with 0 indicating no pain and 10 indicating worst imaginable pain.
Neck pain and disability | At baseline and post-intervention
  Neck Disability Index (NDI) will be used to assess how neck pain affects a patient's daily life and to assess the self-rated disability. A total score is 50, which a higher score indicates a higher disability.
Anxiety and depression | At baseline and post-intervention
  The symptoms of anxiety and depression will be assessed using Hospital Anxiety and Depression Scale (HADS). It includes two subscales: anxiety (HADS-A) and depression (HADS-D). A total score for each subscale ranges from 0 to 21, with higher scores indicating worse symptoms.
Cervical range of motion | At baseline and post-intervention
  Cervical range of motion (degrees) will be measured in flexion, extension, left-right lateral flexion and left-right rotation.
Cervical muscle strength | At baseline and post-intervention
  Cervical muscle strength will be measured in a craniocervical flexion action, using a handheld dynamometer (Newtons).
White matter integrity: fractional anisotropy (FA) and mean diffusivity (MD) | At baseline and post-intervention
  White matter in the brain will be quantified using diffusion tensor imaging (DTI) technique.

CONTACTS AND LOCATIONS:
Overall Officials: Sureeporn Uthaikhup, PhD., Principal Investigator — Department of physical therapy, Chiang Mai university
Locations (1):
- Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jull G, Falla D, Treleaven J, O'Leary S. Management of neck pain disorders: a research informed approach. Edinburgh: Elseiver Limited; 2019.
- [Background] Johnston V, O'Leary S, Comans T, Straker L, Melloh M, Khan A, Sjogaard G. A workplace exercise versus health promotion intervention to prevent and reduce the economic and personal burden of non-specific neck pain in office personnel: protocol of a cluster-randomised controlled trial. J Physiother. 2014 Dec;60(4):233; discussion 233. doi: 10.1016/j.jphys.2014.08.007. Epub 2014 Oct 11. PMID 25306220
- [Background] Sremakaew M, Jull G, Treleaven J, Barbero M, Falla D, Uthaikhup S. Effects of local treatment with and without sensorimotor and balance exercise in individuals with neck pain: protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2018 Feb 13;19(1):48. doi: 10.1186/s12891-018-1964-3. PMID 29433500
- [Background] Maitland GD, Hengeveld E, Banks K, Anglaise K. Vertebral manipulation. 7th ed. Oxford: Butterworth-Heinemann: Elsevier; 2005.
- [Background] de Zoete RMJ, Stanwell P, Weber KA, Snodgrass SJ. Differences in Structural Brain Characteristics Between Individuals with Chronic Nonspecific Neck Pain and Asymptomatic Controls: A Case-Control Study. J Pain Res. 2022 Feb 18;15:521-531. doi: 10.2147/JPR.S345365. eCollection 2022. PMID 35210851
- [Background] Coppieters I, De Pauw R, Caeyenberghs K, Lenoir D, DeBlaere K, Genbrugge E, Meeus M, Cagnie B. Differences in white matter structure and cortical thickness between patients with traumatic and idiopathic chronic neck pain: Associations with cognition and pain modulation? Hum Brain Mapp. 2018 Apr;39(4):1721-1742. doi: 10.1002/hbm.23947. Epub 2018 Jan 11. PMID 29327392
- [Background] Didehdar D, Kamali F, Yoosefinejad AK, Lotfi M. The effect of spinal manipulation on brain neurometabolites in chronic nonspecific low back pain patients: a randomized clinical trial. Ir J Med Sci. 2020 May;189(2):543-550. doi: 10.1007/s11845-019-02140-2. Epub 2019 Nov 26. PMID 31773541
- [Derived] Chaikla R, Sremakaew M, Kothan S, Saekho S, Wantanajittikul K, Uthaikhup S. Effects of manual therapy combined with therapeutic exercise versus routine physical therapy on brain biomarkers in patients with chronic non-specific neck pain in Thailand: a study protocol for a single-blinded randomised controlled trial. BMJ Open. 2023 Apr 24;13(4):e072624. doi: 10.1136/bmjopen-2023-072624. PMID 37094892